CLINICAL TRIAL: NCT06698055
Title: KidREx - Muscle Adaptations in Children and Adults Following a Twelve-week of Resistance Exercise Period Using Either Flywheel or Traditional Weight Stack Devices - a Randomized Controlled Study
Brief Title: Muscle Adaptations in Children and Adults Following Twelve Weeks of Flywheel or Weight Stack Resistance Exercise
Acronym: KidREx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Björn Alkner (Other Government)
Collaborators: Karolinska Institutet (Other); Umeå University (Other); Medical Research Council of Southeast Sweden (Other Government); Swedish Research Council for Sport Science (Other); Linkoeping University (Other Government); The Swedish Research Council (Other Government)
Responsible Party: Sponsor-Investigator, Björn Alkner, Principal Investigator, MD, PhD, Associate professor, Region Jönköping County
Organization: Region Jönköping County (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: RJonkopingC KidREx
Record Dates: First submitted 2023-05-29; First posted 2024-11-20 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-04

CONDITIONS: Resistance Exercise; Muscle Hypertrophy; Skeletal Muscle; EMG; Magnetic Resonance Imaging; Growth Plate Early Closing; Children, Adult
Keywords: Skeletal Muscle; Resistance Exercise; Magnetic Resonance Imaging; EMG; Muscle Hypertrophy; Flywheel Training; Strength Training in Children and Adolescents; Growth Plate; Muscle Adaptation; Muscle Memory; Histology; Immunohistochemistry; Transcriptomics; Methylomics; Proteomics; Functional Outcomes; Physical Activity Monitoring; Physical Self Esteem

STUDY DESIGN:
Intervention Model Description: Randomized controlled resistance exercise intervention study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- aFW = Flywheel resistance exercise intervention group adults (Active Comparator): FW undergo a twelve-week training intervention with alternating two to three sessions per week. At each training session the participant will perform four sets of leg press and a leg extension with seven repetitions per set in each machine were resistance is provided by a flywheel and a weight stack respectively.
  Interventions: Other: Flywheel Resistance Exercise
- aWS = Weight stack resistance exercise intervention group adults (Active Comparator): WS undergo a twelve-week training intervention with alternating two to three sessions per week. At each training session the participant will perform four sets of leg press and a leg extension with seven repetitions per set in each machine were resistance is provided by a flywheel and a weight stack respectively.
  Interventions: Other: Weight Stack Resistance Exercise
- aCON = Control group adults (No Intervention): The CON group will continue living as normally with the aim of remaining at a constant activity level like that at baseline. All groups undergo a baseline test battery witch is repeated following the end of the training period. After the training period all groups enter in to a detraining period were no weight training of the lower limb will be conducted for eight weeks. Following the detraining period the test battery will once more be repeated.
- cFW = Flywheel resistance exercise intervention group children (Active Comparator): FW undergo a twelve-week training intervention with alternating two to three sessions per week. At each training session the participant will perform four sets of leg press and a leg extension with seven repetitions per set in each machine were resistance is provided by a flywheel and a weight stack respectively.
  Interventions: Other: Flywheel Resistance Exercise
- cWS = Weight stack resistance exercise intervention group children (Active Comparator): WS undergo a twelve-week training intervention with alternating two to three sessions per week. At each training session the participant will perform four sets of leg press and a leg extension with seven repetitions per set in each machine were resistance is provided by a flywheel and a weight stack respectively.
  Interventions: Other: Weight Stack Resistance Exercise
- cCON = Control group children (No Intervention): The CON group will continue living as normally with the aim of remaining at a constant activity level like that at baseline. All groups undergo a baseline test battery witch is repeated following the end of the training period. After the training period all groups enter in to a detraining period were no weight training of the lower limb will be conducted for eight weeks. Following the detraining period the test battery will once more be repeated.

INTERVENTIONS:
Other: Flywheel Resistance Exercise — FW is conducted in a leg extension machine (LegExx, Exxentric, Stockholm, Sweden) and leg press machine (YoYo™ Leg Press, nHANCE, Sweden).
  Arms: aFW = Flywheel resistance exercise intervention group adults; cFW = Flywheel resistance exercise intervention group children
Other: Weight Stack Resistance Exercise — WS is conducted in a leg extension machine (Seated leg press, Nordic Gym, Bollnäs, Sweden) and a leg press machine (Seated leg extension, Nordic Gym, Bollnäs, Sweden)
  Arms: aWS = Weight stack resistance exercise intervention group adults; cWS = Weight stack resistance exercise intervention group children

SUMMARY:
The goal of this trial is to compare resistance exercise using traditional techniques and flywheel training to controls in healthy children ages nine to 13 and adults ages 18 to 50. The main questions it aims to answer are:

* The degree of response to resistance exercise in children compared to adults regarding muscle hypertrophy and strength?
* Is there a negative impact on the physis of children due to resistance exercise?

Participants will be randomized to one of three groups, control, traditional resistance exercise, or flywheel. Following a baseline battery of tests, they will enter a 12-week training period, using leg press and leg extension. Additionally, post-training tests are conducted, and an eight-week detraining period commences followed by new tests. Researchers will compare children and adults and each intervention arm to see if children can achieve muscle hypertrophy, the degree and rate of changes in strength, and the potential impact on the physis.

DETAILED DESCRIPTION:
The KidREx-study is an intervention study aiming to investigate the effects of two alternative forms of resistance exercise on adults and children. Exercise forms include leg press and leg extension, in either traditional weight stack machines or flywheel training machines. It has been proposed and discussed that resistance exercise would cause injury to the growth plate and even premature closure of the physis in children. Multiple studies have shown that this is not the case regarding growth height and radiography of the physis. However, the direct effects of resistance exercise on physis using magnetic resonance imaging are yet to be investigated.

This study is a randomized, controlled, prospective intervention study. Two separate groups (children and adults) are included, children ages 9 to 13 and adults ages 18-50. Participants are randomly assigned to one of six arms for the twelve-week intervention period. Arms include two control groups "living as usual" (children and adults), two flywheel training groups (children and adults), and two weight stack training groups (children and adults). Throughout the intervention period, the training groups conduct a total of 30 sessions (alternating between two or three sessions per week). Following the intervention period, all participants enter an 8-week detraining phase, where no organized resistance training is conducted.

At baseline, all participants conduct a test battery including vertical jump height, horizontal jump length, balance tests, and tests of muscle activity in the specific training machines and in an isokinetic dynamometer. In conjunction with the first exercise bout, venous blood samples are obtained from both adults and children, and skeletal muscle biopsies from m. vastus lateralis are obtained from the adults. This procedure is repeated after 12 weeks of training and following the 8-week detraining period. Outcomes related to this, blood samples and muscle tissue, beyond the fiber-specific hypertrophy, will be subject to ancillary studies.

The investigators hypothesize that weight stack training and flywheel training will result in muscle adaptation in both adults and children, where the rate of adaptation is faster for the flywheel training group. Expected muscle adaptation includes an increase in muscle hypertrophy, strength, and functional strength-related outcomes (balance, vertical jump height, and standing long jump). Additionally, the investigators hypothesize that the growth plate of pre- and intra-pubertal children will not be affected negatively by resistance exercise.

ELIGIBILITY:
Inclusion Criteria:

* Adults at the age of 18 to 50 at time of inclusion.
* Children at the age of nine to 13 (attending Swedish middle school) at time of inclusion

Exclusion Criteria:

* Neuromuscular disease.
* Previous or current musculoskeletal injury, primarily of the lower limb, preventing resistance exercise.
* Heavy resistance training of the lower limb at inclusion (i.e., more than one session per week of weight training of the lower limb or other equivalent activity)

Ages: 9 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 91 (Actual)
Dates: Start 2022-08-28 (Actual); Primary Completion 2025-02-02 (Actual); Study Completion 2025-02-12 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Muscle Volume Following 12 Weeks of Resistance Exercies | Time Frame: Before intervention start (0 weeks) and following twelve weeks of training (12 weeks)
  The groups of children and adults will undergo magnetic resonance imaging of the anterior thigh in a standardized fashion. Subsequently, the muscle volume is calculated by contouring cross-sectional area of muscle. Primary analysis is muscle growth of the m. quadriceps femoris in the two active comparator groups compared to the control group.

SECONDARY OUTCOMES:
Changes in muscle thickness | Time Frame: Prior to intervention start, biweekly during the intervention period (i.e., after two, four, six and eight weeks). Additional scans will be performed following the end of intervention (12 weeks) and the end of detraining (20 weeks).
  The group of adults and children undergo ultrasound scans of the anterior thigh in a standardized fashion. The scans will encompass all four heads of the m. quadriceps femoris.
Change from baseline in rate of physeal closure following resistance exercise | Time Frame: Baseline (0 weeks), post training (12 weeks) and post detraining (20 weeks)
  The children will undergo magnetic resonance imaging of the physis of the knee in the non-dominant limb. The degree of closure of the growth plates of the distal femur and proximal tibia will be graded.
Change in muscle volume at 20 weeks | Time Frame: Before intervention start (0 weeks) and end of intervention (12 weeks) compared to volume following the detraining period (20 weeks)]
  The groups of children and adults will undergo magnetic resonance imaging of the anterior thigh in a standardized fashion. Subsequently, the muscle volume (cm3) is calculated by contouring cross-sectional area of muscle. Primary analysis is muscle growth of the m. quadriceps femoris in the two active comparator groups compared to the control group.
Changes in peak torque during isokinetic concentric and eccentric knee extension and flexion | Time Frame: Baseline (0 weeks), post training (12 weeks) and post detraining (20 weeks)
  Concentric and eccentric peak torque (Nm) of the knee extensors and flexors are measured in an Isokinetic dynamometer. Peak torque is measured at 60,120,180 and 300 deg/ sec during concentric actions and 60 deg/sec during eccentric.
Changes in power during isokinetic concentric and eccentric knee extension and flexion | Time Frame: Baseline (0 weeks), post training (12 weeks) and post detraining (20 weeks)
  Concentric and eccentric power (W) of the knee extensors and flexors are measured in an Isokinetic dynamometer. Power is measured at 60,120,180 and 300 deg/ sec during concentric actions and 60 deg/sec during eccentric.
Changes in work during isokinetic concentric and eccentric knee extension and flexion | Time Frame: Baseline (0 weeks), post training (12 weeks) and post detraining (20 weeks)
  Concentric and eccentric work (J) of the knee extensors and flexors are measured in an Isokinetic dynamometer. Work is measured at 60,120,180 and 300 deg/ sec during concentric actions and 60 deg/sec during eccentric.
Changes in muscle activity during isokinetic concentric and eccentric knee extension and flexion measured using sEMG | Time Frame: Baseline (0 weeks), post training (12 weeks) and post detraining (20 weeks)
  Concentric and excentric actions of the knee extensors and flexors are measured in an isokinetic dynamometer using surface electromyography (sEMG) to capture muscle activity from the quadriceps and hamstring musculature. Muscle activity is measured in volts and following post-processing presented in absolute numbers or relative percentages of maximal voluntary contraction (MVC). MVC is acquired during maximal isometric concentric contraction at 60 degrees.
Changes in power during flywheel resistance exercise | Time Frame: Baseline (0 weeks), post training (12 weeks) and post detraining (20 weeks)
  All participants perform test sessions in a flywheel leg press and leg extension where power (W) during the concentric and eccentric face is measured using a rotational encoder.
Changes in muscle activation with flywheel resistance exercise measured using sEMG | Time Frame: Baseline (0 weeks), post training (12 weeks) and post detraining (20 weeks)
  All participants perform test sessions in a flywheel leg press and leg extension where muscle activity of the knee extensors and knee flexors are recorded during two sets and seven repetitions in each machine. Muscle activity (mV) will be adjusted to maximal voluntary contractions (MVC) measured at 90 degrees of knee flexion and extension. Concurrently the joint angel is measured using a goniometer during the entire range of motion.
Changes in power during weight stack resistance exercise | Time Frame: Baseline (0 weeks), post training (12 weeks) and post detraining (20 weeks)
  All participants perform test sessions in a weight stack leg press and leg extension where power (W) during the concentric and eccentric face is measured using a linear encoder.
Changes in muscle activation during weight stack resistance exercise measured using sEMG | Time Frame: Baseline (0 weeks), post training (12 weeks) and post detraining (20 weeks)
  All participants perform test sessions in a weight stack leg press and leg extension where muscle activity of the knee extensors and knee flexors are recorded using electromyography. During two sets and seven repetitions in each machine. Muscle activity (mV) will be adjusted to maximal voluntary contractions (MVC) measured at 90 degrees of knee flexion and extension. Concurrently the joint angel is measured using a goniometer during the entire range of motion.
Changes in power output during training | Time Frame: Continuous power measurements during all training sessions, weeks 1 through 12 weeks
  Power (W) is measured during all training sessions in both training groups. In the flywheel resistance exercise groups using a rotational encoder and in the flywheel stack machine using a linear encoder. Training is performed alternating two to three times weekly during the intervention period.
Changes in Balance | Time Frame: Baseline (0 weeks), post training (12 weeks) and post detraining (20 weeks)
  The participants will perform two standardized sets of tests aimed to quantify their balance, including a series of perturbations and modified-SOT.
Changes in vertical jump height | Time Frame: Baseline (0 weeks), post training (12 weeks) and post detraining (20 weeks)
  The participants will perform two bouts of vertical countermovement jumps, with arms locked upon the hips and with free arms respectively. This will be performed on a force plate and using a motion tracking system.
Changes in isometric maximum strength | Time Frame: Baseline (0 weeks), 2 weeks of intervention, 4 weeks of intervention, 6 weeks of intervention, 8 weeks of intervention and post intervention (12 weeks) and post detraining (20 weeks)
  All participants will perform an isometric maximal contraction of the knee extensors with a 90° knee angle using a force sensor connected in serie with the foot pad in the knee extension weight stack device
Changes in standing long jump | Time Frame: Baseline (0 weeks), 2 weeks of intervention, 4 weeks of intervention, 6 weeks of intervention, 8 weeks of intervention and post intervention (12 weeks) and post detraining (20 weeks)
  The participants will perform three trials of standing long jump. If there is an continues upwards trend, the participants are allowed further trials until a plateau is reached.
Change in type I-fiber cross-sectional area. | Time Frame: Baseline (0 weeks), two weeks of training, six weeks of training, post training (12 weeks) and post detraining (20 weeks).
  Resting muscle biopsies are acquired from the m. vastus laterals muscle of the adults. Fiber-specific staining is performed and cross-sectional area is calculated
Change in type II-fiber cross-sectional area. | Time Frame: Baseline (0 weeks), two weeks of training, six weeks of training, post training (12 weeks) and post detraining (20 weeks).
  Resting muscle biopsies are acquired from the m. vastus laterals muscle of the adults. Fiber-specific staining is performed, and cross-sectional area is calculated
Changes in testosterone levels in children during the intervention | Time Frame: Baseline (0 weeks), post training (12 weeks) and post detraining (20 weeks)
  All child participants will donate blood at baseline, post training and post detraining to assess changes in testosterone (nmol/L) levels.
Changes in estradiol levels in children during the intervention | Time Frame: Baseline (0 weeks), post training (12 weeks) and post detraining (20 weeks)
  All child participants will donate blood at baseline, post training and post detraining to assess changes in estradiol (pmol/L) levels.
Changes in IGF-1 levels in children during the intervention | Time Frame: Baseline (0 weeks), post training (12 weeks) and post detraining (20 weeks)
  All child participants will donate blood at baseline, post training and post detraining to assess changes in insulin-like growth factor 1 (ug/L) levels.
Questionnaire based assessment of physical self-esteem (children) | Time Frame: Baseline (0 weeks), post training (12 weeks) and post detraining (20 weeks)
  Physical self-esteem will be assessed using a translated version (Swedish) of the questionnaire The Children and Youth Physical Self-Perception Profile (CY-PSPP). Total score from 36 to 144 where 144 is the best result.

OTHER OUTCOMES:
Activity level (adults) | Time Frame: Starting one week prior to intervention start and ending one week after detraining time point, a total of 22 weeks.
  Physical activity level will be aggregated to an activity level scored between 0-100, where 0 is the least activity and 100 is the most activity. All participants will wear a smart ring measuring 24h heart rate, accelerometry and pedometry. Data will be aggregated to an activity level using application native software.
Monitoring of physical activity level (children) | All monitors will be worn for one week at three-time points (baseline, 12 weeks, 20 weeks) during the intervention
  All participants will wear accelerometers (wrist and waist) and a smartwatch for heart rate monitoring. Physical activity level will be calculated.
Questionnaire based assessment of physical activity (children) | Baseline (0 weeks), post training (12 weeks) and post detraining (20 weeks)
  Physical will be assessed using a translated version (Swedish) of the questionnaire ASCeND (physical activity scale for children with different abilities).
Hand grip strength | Baseline (0 weeks), post training (12 weeks) and post detraining (20 weeks)
  Hand grip strength will be measured using a dynamometer in both hand at baseline, post-training and detraining.
Readiness score (sleep quality and quantity through adults) | Time Frame: Starting one week prior to intervention start and ending one g week after detraining time point, a total of 22 weeks.
  A readiness score (1-100) based on different parameters. All participants will wear a smart ring measuring 24h heart rate, accelerometry and pedometry. The analysis will include sleep quality, and application native software will be utilized to provide a measurement of sleep quality and quantity combined to one aggregate measure described readiness score.
Monitoring of sleep quality and quantity (children) | All monitors will be worn for one week at three-time points (baseline, 12 weeks, 20 weeks) during the intervention
  An aggregate outcome based on acceleometer data regarding sleep quality and quantity. All child participants will wear accelerometers (wrist and waist).

CONTACTS AND LOCATIONS:
Overall Officials: Björn A Alkner, MD, PhD, Principal Investigator — Department of Orthopaedic Surgery, Eksjö, Region Jönköping County and Department of Biomedical and Clinical Sciences, Linköping University, Linköping, Sweden
Locations (1):
- Department of Orthopaedic Surgery, Höglandssjukhuset District Hospital Eksjö, Eksjö, Region Jönköping County, Sweden

IPD SHARING:
Plan to Share IPD: Yes
All data will be shared upon reasonable request when the data set is is complete
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Upon study completion
Access Criteria: Upon reasonable request